CLINICAL TRIAL: NCT07002385
Title: A Tripartite Biopsychosocial Intervention Program Enhances Mental Health and Quality of Life in Elderly Patients With Depression Secondary to Geriatric Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Seventh People's Hospital (Other Government)
Responsible Party: Principal Investigator, Yan Chen, Principal Investigator, Wenzhou Seventh People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. 20211115
Record Dates: First submitted 2025-05-18; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2022-01

CONDITIONS: Depression Anxiety Disorder; Geriatric Diseases; Mental Health and Quality of Life in Elderly Patients
MeSH Terms: conditions — Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): the control group received standard psychiatric care
- intervention group (Experimental): The intervention group received a biopsychosocial integrated program
  Interventions: Behavioral: control group; Combination Product: Intervention group

INTERVENTIONS:
Behavioral: control group — The control group received standard psychiatric care, which involved physician-led management following clinical guidelines for geriatric disease treatment, including routine medication prescriptions based on diagnostic results. At diagnosis, healthcare providers informed caregivers about the confirmed disease entity, clinical status, and necessary precautionary measures. Monthly mental health lectures were conducted for all patients, covering topics such as common psychological symptoms and coping strategies. Post-discharge, monthly outpatient follow-ups included blood pressure and glucose monitoring. Medication dosages were adjusted if patients reported changes in somatic symptoms.
  Arms: intervention group
Combination Product: Intervention group — The intervention group received a structured biopsychosocial program delivered by a multidisciplinary team. Geriatricians adjusted medications biweekly; rehabilitation therapists led Baduanjin sessions and monitored daily exercises via smart wristbands. Nurses provided CBT-I manuals, and psychologists offered weekly video support. Psychological care included biweekly mindfulness sessions and daily app-guided exercises, with monthly life review activities. Social support involved community events, volunteer roles, and weekly caregiver workshops. Adherence (≥70%) was tracked via app; non-compliance triggered reminders and tailored support. Exercise intensity was regulated by heart rate; patients with ≥5-point HAMD-17 increases were referred. Monthly reviews ensured ongoing quality improvement.
  Arms: intervention group

SUMMARY:
The biopsychosocial integrated intervention program is an effective model for improving holistic health in elderly patients with geriatric disease-related secondary depression, significantly alleviating depressive symptoms, enhancing mental health, and elevating quality of life.

DETAILED DESCRIPTION:
To investigate the effects of a tripartite biopsychosocial intervention program on mental health and quality of life in elderly patients with depression secondary to geriatric diseases. A cluster randomized controlled trial was conducted with 166 elderly patients with secondary depression in our hospital between January 2022 and January 2025. Wards were randomized into an intervention group (n = 83) and a control group (n = 83) using SPSS-generated random sequences. The intervention group received a biopsychosocial integrated program, while the control group received standard psychiatric care. Outcomes were assessed at baseline, 1, 2, and 3 months post-intervention using the 17-item Hamilton Rating Scale for Depression (HAMD-17), mental health indicators [Profile of Mood States (POMS), Five Facet Mindfulness Questionnaire (FFMQ), and Mental Health Continuum-Short Form (MHC-SF)], and the Generic Quality of Life Inventory-74 (GQOLI-74). Patient satisfaction was evaluated post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of depression secondary to geriatric disease (ICD-10 criteria)

Age ≥60 years

Baseline HAMD-17 score ≥14 (mild depression or worse)

Mini-Mental State Examination (MMSE) score ≥24 (no significant cognitive impairment)

Willing and able to provide informed consent (patient or guardian)

Stable on current medications for ≥4 weeks prior to enrollment

Exclusion Criteria:

Primary psychiatric disorders:

Schizophrenia or bipolar disorder

Severe personality disorders

Active suicidal ideation or psychotic symptoms

Recent treatment history:

Antipsychotic medication within 3 months

Electroconvulsive therapy within 6 months

Participation in other interventional trials

Neurological conditions:

Alzheimer's disease or vascular dementia

Parkinson's disease with cognitive impairment

Brain tumors or traumatic brain injury

Medical comorbidities:

Terminal illness with life expectancy <6 months

Uncontrolled cardiovascular disease

Severe hepatic/renal insufficiency (GFR <30 mL/min)

Substance abuse disorders (alcohol or drugs within past year)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Change in Depressive Symptoms Measured by the Hamilton Rating Scale for Depression (HAMD-17) | Baseline, 1 month, 2 months, and 3 months post-intervention.
  The HAMD-17 is a 17-item clinician-administered scale assessing depressive symptom severity (range: 0-52). Higher scores indicate worse depression. Primary outcome: change in HAMD-17 scores from baseline to 3 months post-intervention.

SECONDARY OUTCOMES:
Mental Health Status (Profile of Mood States, POMS) | Baseline, 1 month, 2 months, and 3 months post-intervention.
  The POMS assesses mood disturbances across 40 items (score range: 0-200). Lower scores indicate better mood.
Mindfulness Skills (Five Facet Mindfulness Questionnaire, FFMQ) | Baseline, 1 month, 2 months, and 3 months post-intervention.
  The FFMQ measures mindfulness across 5 facets (score range: 39-195). Higher scores reflect greater mindfulness.
Psychological Well-Being (Mental Health Continuum-Short Form, MHC-SF) | Baseline, 1 month, 2 months, and 3 months post-intervention.
  The MHC-SF evaluates emotional, psychological, and social well-being (score range: 14-70). Higher scores denote better mental health.

OTHER OUTCOMES:
Percentage of Completed Mindfulness Sessions (Per Five Facet Mindfulness Questionnaire Guidelines | Weekly monitoring over 3-month intervention.
  Proportion of attended mindfulness sessions (twice-weekly group sessions + daily APP-guided exercises) out of total prescribed sessions during the 3-month intervention. Adherence threshold: ≥70% (based on FFMQ therapeutic efficacy benchmarks). Data sourced from APP logs and clinician records.
Average Weekly Baduanjin Exercise Duration (Minutes) Tracked via Smart Wristband | Weekly monitoring over 3-month intervention.
  Total minutes of Baduanjin exercise per week, measured via smart wristband synchronization (target: 3×45-minute supervised sessions + 15-20 minutes daily home practice). Heart rate thresholds [(220 - age) × 0.6] ensured safety.
Number of Social Activities Attended (Community/Family Workshops) | Monthly tally over 3-month intervention.
  Count of attended intergenerational activities (monthly) and family workshops (weekly) per participant. Categorized as: 0-25% (low), 26-75% (moderate), or 76-100% (high) of total offered activities.
Change in Morning Salivary Cortisol Concentration (nmol/L) | Baseline and 3 months post-intervention.
  Diurnal cortisol slope measured at awakening (pre- and post-intervention). Collected via passive drool, assayed by ELISA. Reflects HPA axis regulation linked to depression severity.
Change in Serum Brain-Derived Neurotrophic Factor (BDNF) Level (ng/mL) | Baseline and 3 months post-intervention.
  Peripheral BDNF quantified via ELISA from venous blood samples. Explores neurobiological mechanisms of exercise/mindfulness interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Wenzhou Seventh People's Hospital, Wenzhou, Zhejiang, China